CLINICAL TRIAL: NCT01878435
Title: Randomized Controlled Trial of the Impact of Mobile Phone Delivered Reminders and Travel Subsidies to Improve Childhood Immunization Coverage Rates and Timeliness in Western Kenya
Acronym: m-SIMU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Kenya Medical Research Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPP1053900
Record Dates: First submitted 2013-06-10; First posted 2013-06-17 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type b; Measles
Keywords: Short Message System; SMS reminder; mobile phone; cell phone; vaccination; immunization; mHealth
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections; Measles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SMS reminder (Experimental)
  Interventions: Other: SMS reminder
- SMS reminder and Travel subsidy (Experimental)
  Interventions: Other: SMS reminder; Other: Travel subsidy
- Control (No Intervention)
- SMS reminder and Travel subsidy 2 (Experimental)
  Interventions: Other: SMS reminder; Other: Travel subsidy 2

INTERVENTIONS:
Other: SMS reminder
  Arms: SMS reminder; SMS reminder and Travel subsidy; SMS reminder and Travel subsidy 2
Other: Travel subsidy
  Arms: SMS reminder and Travel subsidy
Other: Travel subsidy 2
  Arms: SMS reminder and Travel subsidy 2

SUMMARY:
The project goal is to conduct a randomized controlled trial (RCT) to test whether mobile phone short message system (SMS) reminders, either with or without mobile-phone based travel subsidies will improve timeliness, coverage, and drop-out rates of routine EPI vaccines in rural western Kenya.

ELIGIBILITY:
Inclusion Criteria:

1. Mother of infant aged 0-4 weeks during the study period
2. Current resident of one of the study villages
3. Willing to sign informed consent for the study

Exclusion Criteria:

1. Plans to move out of the study area in the next 6 months
2. Resides in a village with active immunization intervention/program
3. Has already received immunizations other than birth dose of BCG or polio

Ages: 0 Weeks to 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2018 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percent of children immunized | Up to 12 months of age

SECONDARY OUTCOMES:
Percent of fully immunized children (FIC) by study arm | 10 months of age
  FIC = One dose bacille Calmette-Guerin (BCG) vaccine, three doses pentavalent (diphtheria, pertussis, tetanus, hepatitis B, haemophilus influenzae type b) vaccine, three doses polio vaccine and one dose measles vaccine. The proportion of FIC infants by 10 months of age in each of the intervention arms (SMS only and SMS + subsidy) will be separately compared to the control arm using statistical analyses that adjust for the cluster design and any socio-demographic variables that may be unequally distributed across study arms
Proportion of children vaccinated by study arm | Within 2 weeks of each scheduled vaccine date
  The proportion of intervention arm infants that receive vaccination within 2 weeks of the scheduled date will be calculated for each dose of vaccine and compared to the control arm using statistical analyses that adjust for our cluster design and any socio-demographic variables that may be unequally distributed across study arms
Proportion of children dropping out between doses | Age 24 weeks
  Comparison of the differences in percentages of children vaccinated with pentavalent1 and pentavalent3 in the interventions arms compared to this difference in the control arm using statistical analyses that adjust for our cluster design and any socio-demographic variables that may be unequally distributed across study arms
Proportion of children receiving measles and pentavalent vaccines by study arm | Age 24 weeks (pentavalent only), 10 months and age 12 months
  Comparison of vaccine coverage (pentavalent3 and measles, separately) between intervention and control arms
Proportion in each arm vaccinated by mobile phone ownership and by residential distance from a health facility | Age 12 months
  Vaccine coverage analysis stratified by mobile phone ownership and residential distance
Height-for-age,to evaluate if the interventions had impact on other health status indicators | Age 12 months
  Using regression, average height for age in each group will be compared across study groups
Direct costs for each intervention arm | 25 months, approximate time period for deploying interventions
  Costs include SMS messages, the amount of travel subsidy transferred, and the tariffs and fees that are associated with using mobile-money. For each arm, these costs will be divided by the number of children vaccinated and comparisons will be made across study arms
Bed-net usage, to evaluate if the interventions had impact on other indicators of health status | Age 12 months
  Proportion of children using bed-nets will be compared across study groups
Vitamin A coverage, o evaluate if the interventions had impact on other indicators of health status | Age 12 months
  Proportion of children who have received vitamin A supplementation will be compared across study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Gem and Asembo Area, Gem and Asembo Area, Siaya County, Kenya

REFERENCES:
- [Background] Wakadha H, Chandir S, Were EV, Rubin A, Obor D, Levine OS, Gibson DG, Odhiambo F, Laserson KF, Feikin DR. The feasibility of using mobile-phone based SMS reminders and conditional cash transfers to improve timely immunization in rural Kenya. Vaccine. 2013 Jan 30;31(6):987-93. doi: 10.1016/j.vaccine.2012.11.093. Epub 2012 Dec 13. PMID 23246258
- [Background] Gibson DG, Kagucia EW, Ochieng B, Hariharan N, Obor D, Moulton LH, Winch PJ, Levine OS, Odhiambo F, O'Brien KL, Feikin DR. The Mobile Solutions for Immunization (M-SIMU) Trial: A Protocol for a Cluster Randomized Controlled Trial That Assesses the Impact of Mobile Phone Delivered Reminders and Travel Subsidies to Improve Childhood Immunization Coverage Rates and Timeliness in Western Kenya. JMIR Res Protoc. 2016 May 17;5(2):e72. doi: 10.2196/resprot.5030. PMID 27189422
- [Derived] Gibson DG, Ochieng B, Kagucia EW, Were J, Hayford K, Moulton LH, Levine OS, Odhiambo F, O'Brien KL, Feikin DR. Mobile phone-delivered reminders and incentives to improve childhood immunisation coverage and timeliness in Kenya (M-SIMU): a cluster randomised controlled trial. Lancet Glob Health. 2017 Apr;5(4):e428-e438. doi: 10.1016/S2214-109X(17)30072-4. PMID 28288747